CLINICAL TRIAL: NCT04302415
Title: Clinical Study of Metabolomics-based Approach Explore Biomarkers for Metastatic Breast Cancer
Brief Title: Metabolomics Explores Biomarkers for Metastatic Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Zhiyong Yu, Head of Breast surgery, Shandong Cancer Hospital and Institute
Other Study IDs: OMICS Mark
Record Dates: First submitted 2020-03-03; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: metastatic breast cancer; metabolomics; biomarkers; Clinical study
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- only liver metastasis: There is no other intervention, only clinical treatment.
  Interventions: Drug: There is no other intervention, only clinical treatment.
- only lung metastasis: There is no other intervention, only clinical treatment.
  Interventions: Drug: There is no other intervention, only clinical treatment.
- only brain: There is no other intervention, only clinical treatment.
- No distant metastasis: There is no other intervention, only clinical treatment.
  Interventions: Drug: There is no other intervention, only clinical treatment.
- More than two organs metastasis: There is no other intervention, only clinical treatment.

INTERVENTIONS:
Drug: There is no other intervention, only clinical treatment. — There is no other intervention, only clinical treatment.
  Groups: No distant metastasis; only liver metastasis; only lung metastasis

SUMMARY:
RATIONALE: Studying samples of plasm by metabolomics-based approach from women with metastasis breast cancer may help doctors understand the biomarker of visceral metastasis.

PURPOSE: This clinical trial is studying the biomarker of visceral metastasis by metabolomics approach in metastasis breast cancer undergoing treatment.

DETAILED DESCRIPTION:
Imaging evaluation of the effect of chemotherapy on patients with visceral metastases from breast cancer, metabolomics was used to analyze the changes of metabolites in plasma, and to find biomarkers that could reflect visceral metastasis and treatment effects. The purpose is to help clinicians predict whether patients have potential visceral metastases, evaluate the effects of visceral metastasis treatment, and reflect the patient's prognosis.

Patients with visceral metastases on imaging examinations received chemotherapy as planned, and blood samples were collected from patients before and during imaging assessments. Analysis of metabolites in plasma using ultra high performance liquid chromatography. Patient information were collected through medical record, including race, age, height and body mass index, menarche age, menstrual status, menopausal age (if applicable), tobacco and alcohol history, motherhood history, family history, etc.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 yrs.
* Any menopausal status.
* Any hormone receptor status.
* Patients must have histologically or imaging confirmed breast cancer with visceral metastatic.
* Patients must have measurable disease, per RECIST criteria v1.1.21.
* Estimated life expectancy of ≥ 12 weeks.
* Ability to swallow oral medications.
* Participants must have adequate organ function as defined by:

  1. ANC ≥1.5 x 109/L, platelet count ≥100 x 109/L, haemoglobin ≥ 10 g/dL.
  2. creatinine < 1.5 x UNL (upper normal limit).
  3. Total bilirubin < 1.5x UNL.
  4. ALT & AST < 2.5xUNL; alkaline phosphatase < 2.5xUNL.
  5. Creatine phosphokinase (CPK) ≤ 2.5 x UNL.
* Patients with CNS metastatic disease are allowed if the disease is controlled and stable for at least 3 months by CT or MRI.

Exclusion Criteria:

* Current severe, uncontrolled systemic disease (e.g. pulmonary, or metabolic disease; wound healing disorders; ulcers; or bone fractures).
* History of other malignancies.
* No measureable lesion is present, as defined by RECIST 1.1.
* Patients who suffer from a medical or psychiatric condition that, in the opinion of the principal investigator, would impair their ability to participate in the study.
* Concurrent interventional studies.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients must have histologically or imaging confirmed breast cancer with visceral metastatic.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Metabolites changes of plasma by High Performance Liquid Chromatography-Mass Spectrometry (LC-MS). | up to six months
  To assess the changes of metabolites during the process of our observation, and to find out the relationship between metabolite(s) and therapeutic effect.

SECONDARY OUTCOMES:
progression of disease | Up to 10 years
  To observe the duration from the stable condition to progression of disease. Patients were followed up every six months in first five years, then followed up once a year.
overall survival | Up to 10 years
  To observe the duration from the stable condition to death. Patients were followed up every six months in first five years, then followed up once a year.

CONTACTS AND LOCATIONS:
Overall Officials: YU Zhiyong, PhD, Study Chair — Shandong Cancer Hospital and Institute; WANG Fukai, MM, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No